CLINICAL TRIAL: NCT02901847
Title: To Evaluate the Introduction of a Public Health Approach to Peripheral Arterial Disease (PAD) Using National Centre for Sport and Exercise Medicine Facilities.
Acronym: PodPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STH19410
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): PAD tailored care
  Interventions: Other: PAD tailored care

INTERVENTIONS:
Other: PAD tailored care — PAD tailored care

SUMMARY:
The aim of the project is to investigate the clinical and patient centred outcomes of people with Peripheral Arterial Disease (PAD) attending a podiatry led integrated care pathway, utilising advice on diet, activity and smoking cessation. The podiatry clinic will be delivered from the Move More centre (NCSEM) and participants will be encouraged to access these facilities as part of their activity programme which will be agreed with the physical activity team. Primary and secondary outcomes will be clinical - claudication pain, distance walked at 3 and 6 months, blood pressure and lipid monitoring, weight management, reduced BMI, and the success of any smoking cessation. Quality of life and patient satisfaction with the programme will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. adult patient between the ages of 50-90 years,
2. Patient attending for podiatry treatment
3. diagnosis of PAD or is showing signs of symptoms of PAD
4. wishes to take part in the study.

Exclusion Criteria:

1. Anyone unable to give informed consent due to lack of mental capacity.
2. Anyone who would be unable to participate in increased activity due to other co-morbidities

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Distance walked before onset of intermittent claudication | 6 months
  Distance walked before onset of intermittent claudication

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No